CLINICAL TRIAL: NCT06038877
Title: Opinions and Representations of Advanced Practice Nurses (IPA) in Nephrology in France on Clinical Research
Acronym: EBIpa
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN922022/CHUSTE
Record Dates: First submitted 2023-08-29; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Caregivers
Keywords: Advanced practice nurse; Clinical research
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Nephrology Practice Nurses: Advanced Nephrology Practice Nurses in France will be included.
  Interventions: Other: Interviews; Other: Qualitative analysis

INTERVENTIONS:
Other: Interviews — Individual semi-structured interviews
Other: Qualitative analysis — Thematic analysis of the content of responses

SUMMARY:
This single-center study will identify the representations and opinions of Advanced Practise Nurses (IPA) in nephrology in the Auvergne Rhône Alpes (AURA) region about clinical research. The study will consist of individual semi-directive interviews with Advanced Practise Nurses (IPA).

ELIGIBILITY:
Inclusion Criteria:

* Hold a state diploma in advanced practice nursing
* Have been working at the health facilities for at least 3 months
* Working in France

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Advanced Practice Nurses in nephrology in France
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Speeches collected during semi-structured interviews | 5 months
  To explore the beliefs and attitudes of IPA in nephrology about clinical research.

SECONDARY OUTCOMES:
Evaluation of the responses to the follow-up questions | 5 months
  To identify barriers and facilitators of the involvement of this profession in clinical research.

CONTACTS AND LOCATIONS:
Overall Officials: Marion BONJEAN, nurse, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No